CLINICAL TRIAL: NCT00016042
Title: Interleukin 12-Primed Activated T Cells For Patients With Metastatic Renal Cell Carcinoma Or Colorectal Carcinoma (Phase I)
Brief Title: Fluorouracil and Biological Therapy in Treating Patients With Metastatic Kidney or Colorectal Cancer
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: St. Luke's Medical Center (Other)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000068588; STLMC-IMM-0001; NCI-V01-1656
Record Dates: First submitted 2001-05-06; First posted 2004-04-05 (Estimated); Last update posted 2013-09-20 (Estimated); Status verified 2001-10

CONDITIONS: Colorectal Cancer; Kidney Cancer
Keywords: stage IV colon cancer; stage IV rectal cancer; recurrent colon cancer; recurrent rectal cancer; stage IV renal cell cancer; recurrent renal cell cancer
MeSH Terms: conditions — Colorectal Neoplasms; Kidney Neoplasms; Colonic Neoplasms; Rectal Neoplasms; Carcinoma, Renal Cell | interventions — Interferon-alpha; sargramostim; Fluorouracil

INTERVENTIONS:
Biological: lymphokine-activated killer cells
Biological: recombinant interferon alfa
Biological: sargramostim
Drug: fluorouracil

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Biological therapies use different ways to stimulate the immune system and stop cancer cells from growing. Combining chemotherapy with biological therapy may kill more tumor cells.

PURPOSE: Phase I trial to study the effectiveness of fluorouracil combined with biological therapy in treating patients who have metastatic kidney or colorectal cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the safety of fluorouracil and interleukin-12-primed activated T cells (12ATC) with sargramostim (GM-CSF) and interferon alfa in patients with metastatic renal cell cancer or colorectal cancer. II. Determine the maximum tolerated dose of 12ATC in this patient population. III. Determine the clinical response of patients treated with this regimen.

OUTLINE: This is a dose-escalation study of interleukin-12-primed activated T cells (12ATC). Patients receive sargramostim (GM-CSF) subcutaneously (SC) on days 1-5 and undergo leukopheresis on day 6 to obtain peripheral blood mononuclear cells (PBMC). Patients treated at dose level 3 also undergo leukopheresis on day 7. The PBMC are treated with monoclonal antibody anti-CD3, interleukin-12 and interleukin-2 to form 12ATC. Patients receive chemo/immunotherapy comprising fluorouracil IV continuously over 24 hours on day 13 and GM-CSF and interferon alfa SC on days 17, 19, 21, 24, 26, and 28. Patients receive 12ATC IV over 15-30 minutes on days 31, 34, 38, 41, 45, and 48 and interferon alfa SC on days 35, 42, and 49. Cohorts of 3-6 patients receive escalating doses of 12ATC until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 6 patients experience dose-limiting toxicity. Patients are followed at 2 weeks, every 3 months for 1 year, and then every 6 months for 2 years.

PROJECTED ACCRUAL: A total of 9-18 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed metastatic renal cell carcinoma or colorectal carcinoma Failed prior standard or salvage therapy OR Ineligible for standard therapy due to concurrent illness OR Declined standard therapy Bidimensionally measurable disease (by CT scan or MRI) outside prior irradiation port unless documented disease progression after radiotherapy No untreated or unstable treated brain metastasis

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0-2 Life expectancy: More than 3 months Hematopoietic: WBC at least 4,000/mm3 Platelet count at least 100,000/mm3 Total granulocyte count at least 2,000/mm3 Hemoglobin at least 10 g/dL No coagulation disorders such as thrombophlebitis Hepatic: Bilirubin no greater than 2.5 mg/dL SGOT/SGPT less than 3 times upper limit of normal (ULN) Alkaline phosphatase less than 3 times ULN PT/PTT no greater than 1.5 times control Hepatitis B surface antigen negative Renal: Creatinine no greater than 2.0 mg/dL Cardiovascular: No active ischemia and/or ejection fraction less than 45% No unstable angina No uncontrolled congestive heart failure Pulmonary: FEV1 or FVC greater than 65% of predicted No uncontrolled pulmonary embolism Other: No other prior malignancy within the past 5 years except resected basal cell carcinoma or carcinoma in situ of the cervix No active systemic infection No autoimmune disease No uncontrolled thyroid abnormalities No other major medical illness HIV negative Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY: See Disease Characteristics Biologic therapy: More than 1 month since prior biologic therapy or immunotherapy Chemotherapy: More than 1 month since prior chemotherapy (6 weeks for nitrosoureas or mitomycin) Endocrine therapy: At least 4 weeks since prior steroid therapy or steroid-containing compounds At least 2 weeks since prior topical or inhaled steroids No concurrent steroids Radiotherapy: More than 1 month since prior radiotherapy, interstitial brachytherapy, or radiosurgery Surgery: Not specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2001-01

CONTACTS AND LOCATIONS:
Overall Officials: John P. Hanson, MD, Study Chair — St. Luke's Medical Center
Locations (1):
- St. Luke's Medical Center, Milwaukee, Wisconsin, United States